CLINICAL TRIAL: NCT05251259
Title: A Phase 2a, Randomised, Double-Blind, Placebo-Controlled Study to Assess Efficacy and Safety of Atuliflapon Given Orally Once Daily for Twelve Weeks in Adults With Moderate to Severe Uncontrolled Asthma
Brief Title: Study to Assess the Efficacy and Safety of Atuliflapon in Moderate-to-Severe Uncontrolled Asthma
Acronym: FLASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D7552C00001; 2023-509243-27-00 (Other: EU CT Number); 2021-003338-35 (EudraCT Number)
Record Dates: First submitted 2021-12-20; First posted 2022-02-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Efficacy; Safety; Multiple Dose Levels; Adults
MeSH Terms: conditions — Asthma | interventions — AZD5718

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lead-in PK cohort (Atuliflapon) (Experimental): Randomised participants will receive Atuliflapon in Lead-in PK period of the study.
  Interventions: Drug: Atuliflapon
- Lead-in PK cohort (Placebo) (Placebo Comparator): Randomised participants will receive matching placebo to Atuliflapon in Lead-in PK cohort of the study.
  Interventions: Drug: Placebo
- Part 1 (Atuliflapon) (Experimental): Randomised participants will receive Atuliflapon in Part 1 of the study.
  Interventions: Drug: Atuliflapon
- Part 1 (Placebo) (Placebo Comparator): Randomised participants will receive matching placebo to Atuliflapon in Part 1 of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atuliflapon — Randomised participants will receive Atuliflapon
  Other Names: AZD5718
  Arms: Lead-in PK cohort (Atuliflapon); Part 1 (Atuliflapon)
Drug: Placebo — Randomised participants will receive matching placebo to Atuliflapon.
  Arms: Lead-in PK cohort (Placebo); Part 1 (Placebo)

SUMMARY:
This is a randomised, placebo-controlled, double-blind study to assess the efficacy and safety of Atuliflapon administered once daily over a 12-week treatment period to adult participants with moderate to severe uncontrolled asthma.

DETAILED DESCRIPTION:
The study will enroll participants with moderate to severe uncontrolled asthma who are on low-dose inhaled corticosteroid (ICS) - a long-acting beta-agonist (LABA) or medium-to-high-dose ICS with or without LABA background treatment.

The study will be initiated by Lead-in pharmacokinetics (PK) cohort in asthma participants. Participant will be randomised globally, including participants in Lead-in PK cohort (2 arms) and in Part 1 of the study (2 arms).

In the Lead-in PK cohort, participants will be randomised to Atuliflapon or placebo (recruitment completed).

In Part 1 of the study, participants will be stratified by geographical region, and grouped based on high or low levels of biomarker at screening (Visit 1).

ELIGIBILITY:
Inclusion Criteria

Lead-in PK Cohort:

* 18 to 55 years of age inclusive at the time of signing the informed consent at screening Visit 1.
* Bodyweight 50 to 120 kg (inclusive) and BMI 18 to 32 kg/m^2 (inclusive) at screening Visit 1.
* Documented asthma diagnosis ≥12 months prior to screening Visit 1.
* Able to perform acceptable lung function testing for FEV1 according to American Thoracic Society / European Respiratory Society (ATS/ERS) 2019 acceptability criteria.
* Morning pre- bronchodilator (BD) forced expiratory volume (FEV)1 ≥ 40% predicted at screening Visit 1 and Visit 2.
* Treated with low dose inhaled corticosteroid plus long-acting β2-agonist (ICS-LABA) or medium-high dose ICS alone or in combination with LABA at a stable dose for at least 3 months prior to screening Visit 1. Also, treatment with additional asthma controller therapies (eg, LAMA) at a stable dose ≥ 3 months prior to screening Visit 1 is allowed.
* Participant's influenza/pneumonia vaccination is up to date as per local guidelines prior to Visit 2.

General Inclusion Criteria for Part 1:

* Body weight ≥ 40 kg and body mass index (BMI) < 35 kg/m^2.
* Documented history of ≥ 1 severe asthma exacerbation within 1 year prior to screening Visit 1.
* Able to perform acceptable lung function testing for FEV1 according to ATS/ERS 2019 acceptability criteria.
* Morning pre-BD FEV1 between ≥ 40% and ≤ 85% predicted at screening Visit 1 and Visit 3.
* An Asthma Control Questionnaire (ACQ)-6 score ≥ 1.5 at screening Visit 1 and at Visit 3.

Exclusion Criteria

* A severe asthma exacerbation within 8 weeks of screening (visit 1) or within 12 weeks of randomisation (Visit 3).
* A positive test result of an approved antigen test (confirmed by a positive RT-PCR test) or a positive RT-PCR test for SARS-CoV-2, the virus responsible for COVID-19, at screening Visit 1 or at Visit 2 for the PK Lead-in cohort. For Part 1 the testing will be done at Visit 3. Results from the mandatory tests at Visit 2 (PK Lead-in cohort) and Visit 3 (Part 1) must not be older than 48 hours and must be available before randomisation.
* Participants with a significant COVID-19 illness within 6 months of enrolment.
* Clinically important pulmonary disease other than asthma.
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable.
* Any clinically significant cardiac disease.
* History of severe renal disease or history of creatinine clearance < 30 mL/min × m2 calculated using Cockcroft-Gault equation.
* Severe hepatic impairment (Child-Pugh class C).
* Previous hepatotoxicity related to zileuton or leukotriene receptor antagonist (LTRAs) (eg montelukast).
* Participants with a recent history of, or who have a positive test for, infective hepatitis or unexplained jaundice, or participants who have been treated for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Evidence of active tuberculosis (TB), either treated or untreated or latent TB.
* Current or history of alcohol or drug abuse (including marijuana).
* Current diagnosis of cancer, not including in-situ or non-melanoma skin cancer or other previous malignancies where curative therapy was completed at least 5 years prior to screening Visit 1.
* Clinically important ongoing or previous psychiatric disease, especially suicidal behaviour, that in the opinion of the investigator might compromise the safety of the participant in the study.
* Treatment with any serum creatinine-altering drugs within 1 month prior to screening Visit 1 including but not limited to amphotericin, cimetidine, clofibrate, dronedarone, ketoconazole, probenecid, ranolazine, trimethoprim, aminoglycosides, or cephalosporins.
* Treatment with systemic corticosteroid use within 8 weeks (oral) or 12 weeks (intramuscular) before screening (Visit 1) or 12 weeks (oral) or 16 weeks (IM) before randomization (Visit 3).
* Treatment with marketed biologics including benralizumab, mepolizumab, reslizumab, omalizumab, and dupilumab within 6 months of screening Visit 1 or 5 half-lives whichever is longer.
* Treatment with 5-lipoxygenase inhibitors (eg zileuton or other 5-LO inhibiting supplements) within 6 weeks prior to Visit 0 and within 8 weeks prior to Visit 1).Treatment with LTRAs (eg, montelukast) within 2 weeks prior to Visit 0 and within 4 weeks prior to screening Visit 1.
* Inhaled corticosteroid + fast-acting β2 agonist as a reliever (eg Symbicort or Fostair Maintenance and Reliever Treatment) is not allowed 15 days prior to screening Visit 1, during screening (Visit 1)/run-in and the treatment period and preferably 1 week after the last dose of study intervention.
* Live or attenuated vaccines within 4 weeks of screening Visit 1.
* Immunoglobulin or blood products within 4 weeks of screening Visit 1.
* Treatment with Gemfibrozil within 4 weeks of screening Visit 1.
* Any immunotherapy within 6 months of screening Visit 1, except for stable maintenance dose allergen-specific immunotherapy started at least 4 weeks prior to screening Visit 1 and expected to continue through to the end of the follow-up period.
* Potent inducers/inhibitors of cytochrome P450 3A4 within 4 weeks of screening Visit 1.
* Treatment with simvastatin, lovastatin, and atorvastatin at doses > 40 mg per day within 1 month prior to screening Visit 1. Treatment with sensitive cytochrome 3A substrates with narrow therapeutic window should be avoided from randomization to study drug.
* For female participants on ethinyl oestradiol containing combined oral contraceptives, the ethinyl oestradiol doses exceeding 20 mcg per day.
* Concurrent enrolment in another clinical study.
* Previous participation in the current clinical study.
* Participant treated with any investigational drug within 4 months prior to screening Visit 1.
* Known history of allergy or reaction to any component of the study intervention formulation.
* Smokers with smoking history of < 10 pack-years or users of vaping or e-cigarettes, must have stopped at least 6 months prior to screening Visit 1.
* Involvement in the planning and/or conduct of the study.
* Donation of blood (≥ 450 mL) within 3 months or donation of plasma within 14 days before screening Visit 1.
* Major surgery within 8 weeks prior to screening Visit 1, or planned inpatient surgery, major dental procedure or hospitalisation during the screening (Visit 1), treatment or follow-up periods.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Time to first CompEx Asthma event | Baseline up to Week 12
  The clinical efficacy of Atuliflapon Dose A will be assessed by calculating a Hazard Ratio between the treatment arms, Atuliflapon Dose A vs. placebo, in a selected population (based on biomarker level).
  CompEx Asthma, a novel composite endpoint for exacerbations, captures asthma-worsening episodes based on a combination of diary events (worsening in daily peak expiratory flow (PEF), asthma symptoms and reliever medication use) plus severe asthma exacerbation events.

SECONDARY OUTCOMES:
Time to first CompEx Asthma event (Composite endpoint for Exacerbations) | From Baseline up to Week 12
  The clinical efficacy of Atuliflapon Dose A will be identified by determining a selected biomarker threshold using the Hazard Ratio of Atuliflapon Dose A vs. placebo, in all participants (with both high and low levels of biomarker) randomised to either placebo or Atuliflapon arms.
Time to first CompEx Asthma event (Composite endpoint for Exacerbations) | From Baseline up to Week 12
  The clinical efficacy of Atuliflapon Dose A will be assessed using a predetermined biomarker threshold using the Hazard Ratio of Atuliflapon Dose A vs. placebo, in all participants (with both high and low levels of biomarker) randomised to either placebo or Atuliflapon arms.
Change from baseline in Pre-bronchodilator in forced expiratory volume in 1 second (FEV1) | From Baseline up to Week 2, Week 4 and Week 12
  The clinical efficacy of Atuliflapon will be evaluated in comparison to placebo (based on biomarker) of adult participants with moderate-to-severe uncontrolled asthma.
Change from baseline in St. George's Respiratory Questionnaire | From Baseline up to Week 4 and Week 12
  The clinical efficacy of Atuliflapon will be evaluated in comparison to placebo in adult participants with moderate-to-severe uncontrolled asthma.
  The St. George's Respiratory Questionnaire (SGRQ) is a 50-item PRO (Patient Reported Outcomes) instrument to measure the health status of participants with airway obstruction diseases. The questionnaire is divided into two parts: part one consists of 8 items pertaining to the severity of respiratory symptoms in the preceding 4 weeks; part 2 consists of 42 items related to the daily activity and psychosocial impacts of the individual's respiratory condition. The SGRQ yields a total score and three domain scores (symptoms, activity, and impacts). The total score indicates the impact of disease on overall health status. This total score is expressed as a percentage of overall impairment, in which 100 represents the worst possible health status and 0 indicates the best possible health status.
Change from baseline in Asthma Control Questionnaire 6 | From Baseline up to Week 4, Week 8, Week 12
  The clinical efficacy of Atuliflapon will be evaluated in comparison to placebo in adult participants with moderate-to-severe uncontrolled asthma.
  The Asthma Control Questionnaire 6 (ACQ-6) has 6 questions (the top scoring 5 symptoms and daily rescue bronchodilator use). The symptom and bronchodilator use questions on a 7-point scale (0 = no impairment, 6 = maximum impairment). Score 0 means totally controlled and 6 reflects severely uncontrolled.
Change from baseline in average morning and evening Peak Expiratory Flow Measurement | From Baseline up to Week 4, Week 8, Week 12
  The clinical efficacy of Atuliflapon will be evaluated in comparison to placebo in adult participants with moderate-to-severe uncontrolled asthma.
Change from baseline in Daily asthma symptom score (total, daytime, and night-time) | From Baseline up to Week 4, Week 8, Week 12
  The clinical efficacy of Atuliflapon will be evaluated in comparison to placebo in adult participants with moderate-to-severe uncontrolled asthma.
  Asthma symptom scores during night-time and day-time will be assessed by the participant each morning and evening according to the following scoring system: (0) You have no asthma symptoms; (1): You are aware of your asthma symptoms, but you can easily tolerate the symptoms; (2): Your asthma is causing you enough discomfort to cause problems with normal activities (or with sleep); (3): You are unable to do your normal activities (or to sleep) because of your asthma. Here, low score reflects no asthma symptoms and high score suggests severe or frequent symptoms.
Time to first severe asthma exacerbation | From Baseline up to Week 12
  The clinical efficacy of Atuliflapon will be evaluated in comparison to placebo in adult participants with moderate-to-severe uncontrolled asthma. The summary measure for the time-to-event endpoints is being presented as a hazard ratio.
Event status (CompEx Asthma event yes/no) | From Baseline up to Week 12
  The clinical efficacy of Atuliflapon will be evaluated in comparison to placebo in adult participants with moderate-to-severe uncontrolled asthma. The summary measure for the time-to-event endpoints is being presented as a hazard ratio.
Lead-in PK: Area under the curve (AUC) | Day 1 and Day 15
  PK parameter of Atuliflapon will be assessed. Participants will be randomised to Atuliflapon Dose A in the Lead-in PK Cohort.
Lead-in PK: Maximum (or peak) serum concentration (Cmax) | Day 1 and Day 15
  PK parameter of Atuliflapon will be assessed. Participants will be randomised to Atuliflapon Dose A in the Lead-in PK Cohort.
Lead-in PK cohort: Pre-dose trough concentration (Ctrough) | Day 15
  PK parameter of Atuliflapon will be assessed. Participants will be randomised to Atuliflapon Dose A in the Lead-in PK Cohort.
Part 1 Cohort: Atuliflapon plasma concentrations in all participants, pre-dose samples | Baseline, Week 4 and Week 12
  The pre-dose plasma concentrations of Atuliflapon will be summarised.
Number of participants with adverse events (AEs) | Baseline up to Week 12
  The safety and tolerability of Atuliflapon will be assessed in adult participants with moderate-to-severe uncontrolled asthma.

CONTACTS AND LOCATIONS:
Locations (192):
- United States (55):
  - Research Site, Birmingham, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Fountain Valley, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, San Jose, California
  - Research Site, Valencia, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Cutler Bay, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Fayetteville, Georgia
  - Research Site, Lithonia, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Lexington, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Oxon Hill, Maryland
  - Research Site, New Bedford, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, East Orange, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, The Bronx, New York
  - Research Site, Valhalla, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Blue Ash, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Bellaire, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Tomball, Texas
  - Research Site, Milwaukee, Wisconsin
- Argentina (21):
  - Research Site, Bahía Blanca
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Capital Federal
  - Research Site, Ciudad Capital
  - Research Site, Ciudad de Buenos Aire
  - Research Site, Concepción del Uruguay
  - Research Site, Córdoba
  - Research Site, Florida
  - Research Site, Godoy Cruz
  - Research Site, La Plata
  - Research Site, Lobos
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Pilar
  - Research Site, Quilmes
  - Research Site, Ramos Mejía
  - Research Site, Rosario
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Australia (2):
  - Research Site, Adelaide
  - Research Site, Clayton
- Bulgaria (9):
  - Research Site, Kozloduy
  - Research Site, Montana
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Velingrad
  - Research Site, Vidin
- Chile (6):
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Temuco
  - Research Site, Viña del Mar
  - Research Site, Vitacura
- Croatia (5):
  - Research Site, Klenovnik
  - Research Site, Petrinja
  - Research Site, Rijeka
  - Research Site, Split
  - Research Site, Zagreb
- Germany (5):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Marburg
- Hungary (5):
  - Research Site, Gödöllő
  - Research Site, Gyula
  - Research Site, Hajdúnánás
  - Research Site, Pécs
  - Research Site, Szombathely
- Japan (20):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Himeji
  - Research Site, Kawachinagano-shi
  - Research Site, Kobe
  - Research Site, Kodaira-shi
  - Research Site, Koga-shi
  - Research Site, Kokubunji-shi
  - Research Site, Kyoto
  - Research Site, Nakagun
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Setagaya-ku
  - Research Site, Shibuya-Ku
  - Research Site, Tokyo
  - Research Site, Toshima-ku
  - Research Site, Yokohama
- Netherlands (3):
  - Research Site, Breda
  - Research Site, Eindhoven
  - Research Site, Groningen
- Poland (12):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Grudziądz
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Ksawerów
  - Research Site, Lodz
  - Research Site, Ostróda
  - Research Site, Poznan
  - Research Site, Tarnów
  - Research Site, Wroclaw
- Romania (8):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Caracal
  - Research Site, Cluj-Napoca
  - Research Site, Deva
  - Research Site, Iași
  - Research Site, Resca, Com. Dobrosloveni
  - Research Site, Timișoara
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Užice
  - Research Site, Valjevo
- Slovakia (3):
  - Research Site, Levice
  - Research Site, Prešov
  - Research Site, Topoľčany
- South Africa (3):
  - Research Site, Germiston
  - Research Site, Krugersdorp
  - Research Site, Lenasia
- South Korea (4):
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (7):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Benalmádena
  - Research Site, Jerez de la Frontera
  - Research Site, Laredo
  - Research Site, Madrid
  - Research Site, Málaga
- Research Site, Istanbul, Turkey (Türkiye)
- Ukraine (4):
  - Research Site, Chernivtsі
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Vinnytsia
- United Kingdom (16):
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Cardiff
  - Research Site, Chorley
  - Research Site, Corby
  - Research Site, Cottingham
  - Research Site, Glasgow
  - Research Site, Harefield
  - Research Site, Hexham
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Portsmouth
  - Research Site, Reading

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home